CLINICAL TRIAL: NCT05682092
Title: A Randomized Double-blind Controlled Study of Collagen Efficacy on Skin Anti-aging in 30 to 50-Year-Old Women
Brief Title: Study of Collagen Efficacy on Skin Anti-aging in 30 to 50-Year-Old Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Precision Health Food Technology Co. Ltd., (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-SM-11-WL-002
Record Dates: First submitted 2022-12-26; First posted 2023-01-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Skin Laxity; Skin Fold
Keywords: Collagen; skin hydration; skin elasticity; anti-aging
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WonderLab Collagen Tripeptide Drink (Active Comparator): 25ml/bottle, containing the following ingredients per 25ml serving:
  * Collagen 6000 mg
  * Vitamins C 250 mg
  * Hyaluronic acid 50 mg
  * Nicotinamide 0.45 mg
  Interventions: Dietary Supplement: WonderLab Collagen Tripeptide Drink
- Ordinary Drink (Placebo Comparator): 25ml/bottle, containing the following ingredients per 25ml serving:
  * Peach juice 8 mg
  * Erythritol 10 mg
  Interventions: Dietary Supplement: Ordinary Drink

INTERVENTIONS:
Dietary Supplement: WonderLab Collagen Tripeptide Drink — the participant in this arm will use the assigned product 25ml one time, twice a day.
  Arms: WonderLab Collagen Tripeptide Drink
Dietary Supplement: Ordinary Drink — the participant in this arm will use the assigned product 25ml one time, twice a day.
  Arms: Ordinary Drink

SUMMARY:
This goal of this clinical trial is to study the efficacy of collagen supplement on skin moisture and elasticity in middle-aged women of 30-50 years old.

Participants will be assigned two products with and without collagen supplement and use for 2 months, twice a day.

Researchers will compare the two groups whether there are siginificant improvement of skin moisture and elasticity for participants via skin measurement and anaysis system.

DETAILED DESCRIPTION:
This is a two arms, randomized, double-blind controlled trial. Study product plus collagen supplement and placebo product but without collagen will be randomly assigned to 70 eligible participants who will be enrolled at two study sites in Shanghai. Participants need to use the assigned product one bottle (25ml) each time, twice a day and visit the study site for three times (baseline day, day 30 and day 60) during the 2-month study. For each visit, the primary outcomes (skin hydration and skin elasticity) and secondary outcomes (skin barrier, lines/wrinkles, and facial glow,etc.) will be measured with professional equiment and imaging system and recorded to data management system. At the end of the study, the study data will exported and analyzed to validate the assumption that the collagen could improve skin moisture content and elasticity in middle-aged women of 30-50 years old.

ELIGIBILITY:
Inclusion Criteria:

* Chinese females, age between 30-50;
* Be in general good health;
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate;
* Have mild to moderate darker skin tone 3 on Unilever visual scale of 1~9;
* Have mild pigmentation level 2 on Unilever visual scale of 0~9;
* Have visual grading score on crow's feet 3 on Unilever visual scale of 0~9;
* Have visual grading score on peri-oral 3 on Unilever visual scale of 0~9;
* Have visual grading score on nasolabial folds 3 on Unilever visual scale of 0~9;
* Tolerate to well-known anti-aging actives;
* Agree to not use any other creams, lotions, moisturizers on the face, other than what is provided for the duration of the study;
* Agree to refrain from wearing make-up (such as foundation, eye shadow, lipstick etc.) or any skin care products on the face on the study visits;
* Agree to avoid washing the treatment site area for two hours following product application and agree to avoid washing appliances (i.e., sponge, wash cloth, loofah, etc.).

Exclusion Criteria:

* Have used any skin lightening /anti-aging benefits products at least one month before this study
* Subject having done facial injections and/or aesthetic surgery.
* Be involved in any aspect of test administration, i.e., evaluating or overseeing activities related to product.
* Have participated in any clinical study involving the test sites within the previous 6 months, or is subject participating in any clinical study concurrently.
* Have a history of any type of bottlecer, including but not limited to any type of skin bottlecer (squamous or basal cell carcinoma at the treatment site) or history of malignant melanoma at any body site.
* Have a history of skin disease or the presence of a skin condition on the test sites that the Investigator feels would interfere with the study.
* Be taking antihistamines (> 3x/week) or anti-inflammatory (> 8x/week) on a regular basis, or has the subject taken systemic or topical steroidal medications within 4 weeks of study enrolment.
* Have any of the following conditions or factors that the investigator believes may affect the response of the skin or the interpretation of the test results, including, but not limited to, diabetes, pregnancy, lactation.
* Have any cuts/abrasions on the test site at baseline.
* Have had a suspicious skin lesion removed by a dermatologist at any time.
* The subject is an employee of sponsor or the site conducting the study.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — the participants must be middle-aged women of 30-50 years old
Enrollment: 70 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Skin Elasticity | baseline day 0, day 30, day 60
  The changes of skin elasticity by CK Cutometer MPA580
Skin Moisture | baseline day 0, day 30, day 60
  The changes of skin moisture by Corneometer CM 825

SECONDARY OUTCOMES:
Skin Barrier | baseline day 0, day 30, day 60
  The changes of skin barrier in terms of TEWL (Trans Epidermal Water Loss) by Aquaflux F200
Lines/Wrinkles | baseline day 0, day 30, day 60
  The changes of the lines/wrinkles on the face by Miravex Antera 3D imaging system
Skin Diagnosis | baseline day 0, day 30, day 60
  The skin diagnosis (4 modes and 2 side views) with VISIA CR Facial Imaging System

CONTACTS AND LOCATIONS:
Overall Officials: Yun Wang, MD, Principal Investigator — NO. 9 Hospital affiliated to Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Ai'er Hospital, Shanghai, Shanghai Municipality
  - SPRIM Central Lab, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proksch E, Schunck M, Zague V, Segger D, Degwert J, Oesser S. Oral intake of specific bioactive collagen peptides reduces skin wrinkles and increases dermal matrix synthesis. Skin Pharmacol Physiol. 2014;27(3):113-9. doi: 10.1159/000355523. Epub 2013 Dec 24. PMID 24401291
- [Background] Zague V, de Freitas V, da Costa Rosa M, de Castro GA, Jaeger RG, Machado-Santelli GM. Collagen hydrolysate intake increases skin collagen expression and suppresses matrix metalloproteinase 2 activity. J Med Food. 2011 Jun;14(6):618-24. doi: 10.1089/jmf.2010.0085. Epub 2011 Apr 11. PMID 21480801
- [Background] Proksch E, Segger D, Degwert J, Schunck M, Zague V, Oesser S. Oral supplementation of specific collagen peptides has beneficial effects on human skin physiology: a double-blind, placebo-controlled study. Skin Pharmacol Physiol. 2014;27(1):47-55. doi: 10.1159/000351376. Epub 2013 Aug 14. PMID 23949208
- [Background] Nouveau-Richard S, Yang Z, Mac-Mary S, Li L, Bastien P, Tardy I, Bouillon C, Humbert P, de Lacharriere O. Skin ageing: a comparison between Chinese and European populations. A pilot study. J Dermatol Sci. 2005 Dec;40(3):187-93. doi: 10.1016/j.jdermsci.2005.06.006. Epub 2005 Sep 8. PMID 16154324
- [Background] Liang J, Pei X, Zhang Z, Wang N, Wang J, Li Y. The protective effects of long-term oral administration of marine collagen hydrolysate from chum salmon on collagen matrix homeostasis in the chronological aged skin of Sprague-Dawley male rats. J Food Sci. 2010 Oct;75(8):H230-8. doi: 10.1111/j.1750-3841.2010.01782.x. Epub 2010 Sep 24. PMID 21535500